CLINICAL TRIAL: NCT04298177
Title: Personalized Atrial Fibrillation Ablation With the QDOT Catheter - The QDOT-by-LAW Trial
Brief Title: Personalized Atrial Fibrillation Ablation With QDOT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio Berruezo, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Antonio Berruezo, MD, PhD, Research Coordinator of the Heart Institute, Centro Medico Teknon
Organization: Centro Medico Teknon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QDOT-by-LAW
Record Dates: First submitted 2020-02-29; First posted 2020-03-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; pulmonary vein isolation; left atrial wall thickness; high-power short-duration ablation; QDOT
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a two-arm, single-blind, single-center, randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- QDOT-LAWT (Experimental): A QDOT® 3.5-mm open-irrigated contact force-sensing RF ablation catheter (Biosense Webster, Inc., Irvine, CA, USA) will be used.
  The primary ablation mode for PVI will depend on the calculated LAWT at each atrial point, as follows:
  **< 3.5-mm LAWT (red, and yellow colors): vHPSD ablation will be performed. If <1-mm LAWT (red color): Power 90 W; the duration of RF applications will be reduced to 2 seconds. If 1-3.5 mm LAWT (yellow color): Power 90 W; the duration of RF applications will be 4 seconds, according to the QDOT-FAST protocol.
  **> 3.5-mm LAWT (green color): QMODE ablation will be performed. 50 W with AI target = 500
  Interventions: Device: Atrial fibrillation ablation using the QDOT® catheter
- CLOSE (Active Comparator): In the CLOSE arm, the use of MDCT-derived LAWT information will not be available for the operator. A ThermoCool® SmartTouch® 3.5-mm open-irrigated contact force-sensing RF ablation catheter (Biosense Webster, Inc., Diamond Bar, CA, USA) will be used. The ablation will be performed using a proprietary RF generator (SMARTABLATE®; Biosense Webster, Diamond Bar, CA, USA).
  Ablation will be performed according to the CLOSE study settings: Power-controlled mode (without ramping) with 25 to 35 W (irrigation flow 30 ml/min). RF will be delivered until an AI of ≥ 400 at the posterior wall/roof and ≥ 550 at the anterior wall are reached.
  Interventions: Procedure: Standard atrial fibrillation ablation

INTERVENTIONS:
Device: Atrial fibrillation ablation using the QDOT® catheter — Atrial fibrillation ablation will be performed using the QDOT® catheter. The ablation mode will be selected according to the MDCT-derived LAWT information.
  Other Names: Pulmonary vein isolation
  Arms: QDOT-LAWT
Procedure: Standard atrial fibrillation ablation — Atrial fibrillation ablation will be performed using the SmartTouch® catheter. The ablation parameters will be adjusted according to the settings previously described in the CLOSE study.
  Other Names: Pulmonary vein isolation
  Arms: CLOSE

SUMMARY:
Circumferential pulmonary vein isolation (PVI) has become a mainstay in the treatment of atrial fibrillation (AF), particularly in symptomatic patients with paroxysmal AF (PAF) intolerant or refractory to medical treatment. The safety and short-term performance of the novel QDOT® catheter (Biosense Webster, Irvine, CA, USA), that allows for a high-power short-duration (HPSD) ablation, has already been evaluated in the QDOT-FAST clinical study, with favorable data on feasibility and safety, and lowered fluoroscopy and procedure times needed to achieve complete PVI. HPSD ablation was based on immediate heat formation during the resistive phase, affecting a small tissue depth at 90 W/4 s (irrigation at 8 ml/min) with a temperature limit of 65ºC.

However, up to date there are no randomized studies evaluating the real usefulness of the QDOT® catheter. Longer-term follow-up is still required to verify the long-term effectiveness and correlations between short-term follow-up and arrhythmia recurrence when using this catheter. The impact of this novel catheter, when used in conjunction with a personalized ablation protocol that uses the information of left atrial wall thickness (LAWT) to modulate the AI target at each ablation point, compared with a standard ablation protocol following the published CLOSE study criteria is already unknown.

DETAILED DESCRIPTION:
Circumferential pulmonary vein isolation (PVI) has become a mainstay in the treatment of atrial fibrillation (AF), particularly in symptomatic patients with paroxysmal AF (PAF) intolerant or refractory to medical treatment. Dormant conduction and pulmonary vein reconnections are responsible for AF/atrial tachycardia (AT) recurrences owing to incomplete non-transmural ablation lesions that generate gaps on ablation lines.

The advent of contact force (CF) catheters has represented a significant milestone when reaching better efficiency in RF delivery, helping to achieve better PVI rates after AF ablation. The benefits of CF sensing have been already demonstrated in both the SMART AF (THERMOCOOL® SMARTTOUCH® Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation) and the TOCCASTAR (TactiCath® Contact Force Ablation Catheter Study for Atrial Fibrillation) studies. Moreover, CF stability is also an important predictor of reduced arrhythmia recurrence.

Recently, ablation index (AI) (CARTO3® V4; Biosense Webster, Inc, Diamond Bar, CA, USA) was developed as a novel marker of lesion quality that, for the first time, incorporates CF as well as duration, and power delivery. The recent CLOSE clinical study analyzed the utility of ablation index (AI), a novel formula developed to assess real-time effect of RF delivery and improve the rates of permanent PVI, with 91.3% of the patients free from AF/AT/atrial flutter (AFL) at 12 months follow-up. The CLOSE protocol targeted an interlesion distance (ILD) of 6 mm and AI ≥ 400 at the posterior wall and ≥550 at the anterior wall.

However, another recent study revealed that AI, while being very reliable across a range of CF values, may be 'penalized' by small contact angles and high-power RF applications, which could decrease the lesion size at the same AI. The small lesion size at narrow contact angle may be explained by tip temperature drop due to saline flow from irrigation holes located at the side of the catheter tip during RF application. Bourier et al. reported that extremely high-power RF applications (> 50 W) resulted in significantly smaller lesion depth for short-duration applications (n = 120).

In a swine model, high-power short-duration (HPSD) ablation resulted in 100% contiguous lines with all transmural lesions, whereas standard ablation (25 W for 20 s) had linear gaps in 25% and partial thickness lesions in 29%. The authors of this experimental study used a novel ablation catheter that incorporates 6 thermocouples symmetrically embedded in the circumference of the tip electrode, named QDOT® catheter (Biosense Webster, Irvine, CA, USA). This catheter permits to control the confounding effect of the cold irrigation fluid during ablation, while having an improved irrigation system. In the same study, ablation with HPSD produced wider lesions at similar depth, and improved lesion-to-lesion uniformity with comparable safety endpoints. Given the aforesaid, it can be hypothesized that larger diameter of HPSD lesions might contribute to a complete encirclement of PV, by ensuring better contiguity between adjacent lesions, while the reduced lesion depth may still achieve lesion transmurality in atrial tissue, diminishing the risk of collateral tissue damage.

The safety and short-term performance of the QDOT® catheter (Biosense Webster, Irvine, CA, USA) has already been evaluated in the QDOT-FAST clinical study (Clinical Study for Safety and Acute Performance Evaluation of the THERMOCOOL SMARTTOUCH SF-5D System Used With Fast Ablation Mode in Treatment of Patients With Paroxysmal Atrial Fibrillation), with favorable data on feasibility and safety, and lowered fluoroscopy and procedure times needed to achieve complete PVI. HPSD ablation was based on immediate heat formation during the resistive phase, affecting a small tissue depth at 90 W/4 s (irrigation at 8 ml/min) with a temperature limit of 65ºC.

Up to date, there are no randomized studies evaluating the real usefulness of the QDOT® catheter. Moreover, longer-term follow-up is required to verify the long-term effectiveness and correlations between short-term follow-up and arrhythmia recurrence when using this catheter. The impact of the QDOT® catheter, when used in conjunction with a personalized ablation protocol that uses the information of left atrial wall thickness (LAWT) to modulate the AI target at each ablation point, compared with a standard ablation protocol (CLOSE study criteria) is already unknown.

Our research hypothesis is that QDOT-by-LAW, a personalized protocol that uses a dedicated vHPSD catheter, a multichannel radiofrequency (RF) generator with a vHPSD ablation mode, and integrated LAWT information to adapt the ablation index (AI) target to the subjacent LAWT, is safe, while showing at least the same efficacy and better efficiency than the CLOSE protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Indication for paroxysmal atrial fibrillation ablation.
* Signed informed consent

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Previous AF redo procedure.
* Impossibility to perform a pre-procedural CT scan.
* Concomitant investigation treatments.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 1 year
  Survival free of any atrial arrhythmia at the 3-month, 6-month, and 12-month follow-up.

SECONDARY OUTCOMES:
Procedure time | 1 month
  Procedure time (skin to skin)
Radiofrequency time | 1 month
  Radiofrequency time
Number of radiofrequency applications | 1 month
  Number of applications (total/per PVI RF line/per segment)
Fluoroscopy time | 1 month
  Fluoroscopy time
First pass isolation rate | 1 month
  First pass isolation rate
Early PV reconnection rate | 1 month
  Early PV reconnection rate
Incidence of peri-procedural complications | 1 month
  Incidence of peri-procedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Medico Teknon
Locations (1):
- Teknon Medical Center, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Ouyang F, Tilz R, Chun J, Schmidt B, Wissner E, Zerm T, Neven K, Kokturk B, Konstantinidou M, Metzner A, Fuernkranz A, Kuck KH. Long-term results of catheter ablation in paroxysmal atrial fibrillation: lessons from a 5-year follow-up. Circulation. 2010 Dec 7;122(23):2368-77. doi: 10.1161/CIRCULATIONAHA.110.946806. Epub 2010 Nov 22. PMID 21098450
- [Background] Cappato R, Negroni S, Pecora D, Bentivegna S, Lupo PP, Carolei A, Esposito C, Furlanello F, De Ambroggi L. Prospective assessment of late conduction recurrence across radiofrequency lesions producing electrical disconnection at the pulmonary vein ostium in patients with atrial fibrillation. Circulation. 2003 Sep 30;108(13):1599-604. doi: 10.1161/01.CIR.0000091081.19465.F1. Epub 2003 Sep 8. PMID 12963643
- [Background] Kuck KH, Hoffmann BA, Ernst S, Wegscheider K, Treszl A, Metzner A, Eckardt L, Lewalter T, Breithardt G, Willems S; Gap-AF-AFNET 1 Investigators*. Impact of Complete Versus Incomplete Circumferential Lines Around the Pulmonary Veins During Catheter Ablation of Paroxysmal Atrial Fibrillation: Results From the Gap-Atrial Fibrillation-German Atrial Fibrillation Competence Network 1 Trial. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003337. doi: 10.1161/CIRCEP.115.003337. PMID 26763226
- [Background] Natale A, Reddy VY, Monir G, Wilber DJ, Lindsay BD, McElderry HT, Kantipudi C, Mansour MC, Melby DP, Packer DL, Nakagawa H, Zhang B, Stagg RB, Boo LM, Marchlinski FE. Paroxysmal AF catheter ablation with a contact force sensing catheter: results of the prospective, multicenter SMART-AF trial. J Am Coll Cardiol. 2014 Aug 19;64(7):647-56. doi: 10.1016/j.jacc.2014.04.072. PMID 25125294
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733
- [Background] Reddy VY, Pollak S, Lindsay BD, McElderry HT, Natale A, Kantipudi C, Mansour M, Melby DP, Lakkireddy D, Levy T, Izraeli D, Sangli C, Wilber D. Relationship Between Catheter Stability and 12-Month Success After Pulmonary Vein Isolation: A Subanalysis of the SMART-AF Trial. JACC Clin Electrophysiol. 2016 Nov;2(6):691-699. doi: 10.1016/j.jacep.2016.07.014. Epub 2016 Nov 21. PMID 29759747
- [Background] Das M, Loveday JJ, Wynn GJ, Gomes S, Saeed Y, Bonnett LJ, Waktare JEP, Todd DM, Hall MCS, Snowdon RL, Modi S, Gupta D. Ablation index, a novel marker of ablation lesion quality: prediction of pulmonary vein reconnection at repeat electrophysiology study and regional differences in target values. Europace. 2017 May 1;19(5):775-783. doi: 10.1093/europace/euw105. PMID 27247002
- [Background] El Haddad M, Taghji P, Phlips T, Wolf M, Demolder A, Choudhury R, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Determinants of Acute and Late Pulmonary Vein Reconnection in Contact Force-Guided Pulmonary Vein Isolation: Identifying the Weakest Link in the Ablation Chain. Circ Arrhythm Electrophysiol. 2017 Apr;10(4):e004867. doi: 10.1161/CIRCEP.116.004867. PMID 28381417
- [Background] Taghji P, El Haddad M, Phlips T, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Evaluation of a Strategy Aiming to Enclose the Pulmonary Veins With Contiguous and Optimized Radiofrequency Lesions in Paroxysmal Atrial Fibrillation: A Pilot Study. JACC Clin Electrophysiol. 2018 Jan;4(1):99-108. doi: 10.1016/j.jacep.2017.06.023. Epub 2017 Sep 27. PMID 29600792
- [Background] Kawaji T, Hojo S, Kushiyama A, Nakatsuma K, Kaneda K, Kato M, Yokomatsu T, Miki S. Limitations of lesion quality estimated by ablation index: An in vitro study. J Cardiovasc Electrophysiol. 2019 Jun;30(6):926-933. doi: 10.1111/jce.13928. Epub 2019 Apr 2. PMID 30912209
- [Background] Bourier F, Duchateau J, Vlachos K, Lam A, Martin CA, Takigawa M, Kitamura T, Frontera A, Cheniti G, Pambrun T, Klotz N, Denis A, Derval N, Cochet H, Sacher F, Hocini M, Haissaguerre M, Jais P. High-power short-duration versus standard radiofrequency ablation: Insights on lesion metrics. J Cardiovasc Electrophysiol. 2018 Nov;29(11):1570-1575. doi: 10.1111/jce.13724. Epub 2018 Sep 25. PMID 30168230
- [Background] Leshem E, Zilberman I, Tschabrunn CM, Barkagan M, Contreras-Valdes FM, Govari A, Anter E. High-Power and Short-Duration Ablation for Pulmonary Vein Isolation: Biophysical Characterization. JACC Clin Electrophysiol. 2018 Apr;4(4):467-479. doi: 10.1016/j.jacep.2017.11.018. Epub 2018 Feb 2. PMID 30067486
- [Background] Barkagan M, Contreras-Valdes FM, Leshem E, Buxton AE, Nakagawa H, Anter E. High-power and short-duration ablation for pulmonary vein isolation: Safety, efficacy, and long-term durability. J Cardiovasc Electrophysiol. 2018 Sep;29(9):1287-1296. doi: 10.1111/jce.13651. Epub 2018 Jun 20. PMID 29846987
- [Background] Reddy VY, Grimaldi M, De Potter T, Vijgen JM, Bulava A, Duytschaever MF, Martinek M, Natale A, Knecht S, Neuzil P, Purerfellner H. Pulmonary Vein Isolation With Very High Power, Short Duration, Temperature-Controlled Lesions: The QDOT-FAST Trial. JACC Clin Electrophysiol. 2019 Jul;5(7):778-786. doi: 10.1016/j.jacep.2019.04.009. Epub 2019 May 8. PMID 31320006
- [Derived] Falasconi G, Penela D, Soto-Iglesias D, Francia P, Saglietto A, Turturiello D, Viveros D, Bellido A, Alderete J, Zaraket F, Franco-Ocana P, Huguet M, Camara O, Vatasescu R, Ortiz-Perez JT, Marti-Almor J, Berruezo A. Personalized pulmonary vein isolation with very high-power short-duration lesions guided by left atrial wall thickness: the QDOT-by-LAWT randomized trial. Europace. 2024 Mar 30;26(4):euae087. doi: 10.1093/europace/euae087. PMID 38652090